CLINICAL TRIAL: NCT00923104
Title: An Exploratory Evaluation of Biomarkers in Blister Fluid in Healthy Volunteers and Irradiated Skin
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090120; 09-C-0120
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Healthy Volunteer; Prostate Cancer
Keywords: Radiation; Blister; Healthy Volunteer; Samples; Natural History; Prostate Cancer; Breast Cancer; HV
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Blister

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/healthy volunteers: healthy volunteers
- 2/patients: subjects with breast cancer, ductal carcinoma in situ, and adenocarcinoma of prostate

SUMMARY:
Background:

* Blister fluid contains many of the same biomarkers (substances that can be used to determine the effects of certain kinds of treatments) as blood and urine samples, particularly regarding changes in the skin.
* The Radiation Oncology Branch and others are conducting research studies that require blood and urine samples from healthy volunteers and from patients with cancer. In addition to these samples, researchers would like to collect the fluid from blisters to examine markers of inflammation in the skin.

Objectives:

* To compare blood, urine, and blister fluid samples of patients with cancer who are undergoing radiation therapy to that of volunteers without cancer who will not be receiving radiation therapy.
* To gather more information about the effects of radiation therapy on the skin and body fluids of individuals.

Eligibility:

* Patients 18 years of age and older who will be receiving radiation therapy for either breast or prostate cancer.
* A separate group of healthy volunteers will also participate in this study.

Design:

* Physical examination and blood samples to determine eligibility for the study.
* Blister induction, conducted before the start of radiation treatment, at completion of radiotherapy (last day of treatment), and at a visit 12 months after the end of radiation treatment.
* Blisters will be created through the use of a suction blister device on the hip (for patients with prostate cancer) or on the treated breast or location of removed breast (for patients with breast cancer).
* Blisters will take approximately 30 minutes to form, and fluid will be removed with a needle and syringe.
* Blood and urine samples will also be collected at this time.
* Radiation treatment for breast or prostate cancer will be conducted according to standard procedures, or as directed by a separate research protocol.
* Evaluations during the treatment period:
* Physical examination, including vital signs and body weight checks, and pregnancy test for women who can become pregnant.
* Blood and urine tests.
* Disease evaluation.
* Post-treatment evaluations:
* Clinic visits at months 1, 3, 6, 9, and 12 after the end of radiation therapy for physical examination and disease assessment.
* Study will end 1 year after the final radiation treatment, upon the collection of the final (third) blister fluid sample.

DETAILED DESCRIPTION:
BACKGROUND

Blister fluid has been used to measure cytokine expression, proteomic profiles, and pharmacokinetics in a variety of disease states.

Blister fluid inside radiation treatment fields has been shown to have altered expression of cytokines and products of collagen metabolism.

Evaluation of blister fluid in normal skin inside and outside the radiation field may allow the development of a minimally invasive marker of radiation exposure or damage induced by radiation in irradiated skin.

OBJECTIVES

This protocol will evaluate the ability to determine a cytokine pattern and global changes at the protein level measured in blister fluid that correlates with radiation exposure, absorbed skin dose, or skin toxicity from patients receiving radiation.

ELIGIBILITY

Patients in whom radiotherapy is required for standard management of theirbreast or prostate cancer.

Healthy volunteers with no history of cutaneous inflammatory condition of the skin such as eczema, or psoriasis.

DESIGN

This protocol is designed to evaluate blister fluid in and out of the radiation field in patients that are receiving radiation therapy and in healthy volunteers.

Patients will undergo blister induction and blister fluid collection prior to treatment outside of the radiation field, and after completion of radiation within the radiation field.

Blisters will be induced in a non-sun exposed area and if possible in matched sites (i.e. left and right).

ELIGIBILITY:
* ELIGIBILITY CRITERIA

ELIGIBILITY CRITERIA FOR PATIENTS RECEIVING RADIOTHERAPY:

INCLUSION CRITERIA:

1. Histological diagnosis: Pathologically confirmed diagnosis of 1) invasive breast cancer, 2) ductal carcinoma in situ, or 3) adenocarcinoma of the prostate.
2. Patients in whom the management of the histologic diagnosis will include radiation treatment as part of standard clinical management.
3. Patients in whom the extent of disease is considered local or locoregional (i.e. requiring definitive radiotherapy to the breast or prostate).
4. Patients must be older than 18 years of age.
5. Patients must have a primary medical or surgical oncologist in the community or at NCI who is willing to collaborate with the ROB staff in the clinical management of the patient.
6. Patients of childbearing or child- fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated with radiotherapy on this study.
7. Patients must have an ECOG performance status of 0-2 and a life expectancy greater than 12 months.

EXCLUSION CRITERIA:

1. Patients with a history of chronic skin disease such as psoriasis, eczema, or history of keloid formation.
2. Patients requiring concurrent use of topical steroids
3. Patients requiring concurrent use of glucocorticoid therapy.
4. Patients who have received topical or systemic chemotherapy within 4 weeks of enrollment (not including hormonal agents such as antiandrogens, GnRH agonists, aromatase inhibitors, tamoxifen, and similar agents) are excluded.
5. Patients requiring concurrent chemotherapy with radiotherapy except as noted in (Protocol section 2.3.1) are excluded.
6. Patients with a history of lupus erythematosis, scleroderma, ataxia telengiectasia or other known hypersensitivity to therapeutic radiation.
7. Patients with prior radiotherapy to the site which would be used for blister induction.
8. Patients who are pregnant because of the potential mutagenic effects of radiation on a developing fetus or newborn.
9. Patients with unrelated systemic illness which in the judgment of the Principal Investigator (PI) would compromise the patient s ability to tolerate this therapy or are likely to interfere with the study procedures or results.
10. Patients who are in the estimation of the PI, deemed unable or unlikely to adhere to protocol treatment.
11. Patients with significant skin atrophy that would interfere with blister formation.
12. Breast cancer patients in whom the site of radiotherapy includes a myocutaneous flap or skin graft.

ELIGIBILITY CRITERIA FOR HEALTHY VOLUNTEERS:

INCLUSION CRITERIA:

1. Healthy volunteers older than 18 years of age.
2. Ability to provide informed consent.

EXCLUSION CRITERIA:

1. History of chronic skin disease such as psoriasis, eczema, or history of keloid formation.
2. Concurrent use of glucocorticoid therapy.
3. History of lupus erythematosis, scleroderma, ataxia telengiectasia or other known hypersensitivity to therapeutic radiation.
4. Prior radiotherapy to the site which would be used for blister induction (for benign or malignant causes).
5. Unrelated systemic illness which in the judgment of the Principal Investigator (PI) would compromise the patient s ability to tolerate blister induction or are likely to interfere with blister healing, the study procedures, or the study results.
6. Darkly pigmented skin in whom pigmentation changes are a likely complication
7. Significant skin atrophy that would interfere with blister formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in whom radiotherapy is required for standard management of their breast or prostate cancer. Healthy volunteers with no history of cutaneous inflammatory condition of the skin such as eczema, or psoriasis.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2009-04-23 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
To determine if cytokine levels in blister fluid change following exposure of the skin to low or high dose radiation | study completion
  The primary objectives of this study are (i) to determine if cytokine levels in blister fluid change following exposure of skin to low or high dose radiation, and (ii) to compare cytokine levels in blister fluid from unirradiated skin in normal controls, breast cancer patients, and prostate cancer patients. We will examine IL-1 beta, IL6, TNF-alpha, and MMP-1 and -3 for the primary analysis. The remaining cytokines will be examined in secondary analyses.
To compare blister fluid cytokine levels in blister fluid from unirradiated skin in normal controls, breast cancer patients, and prostate cancer patients | study completion
  The primary objectives of this study are (i) to determine if cytokine levels in blister fluid change following exposure of skin to low or high dose radiation, and (ii) to compare cytokine levels in blister fluid from unirradiated skin in normal controls, breast cancer patients, and prostate cancer patients. We will examine IL-1 beta, IL6, TNF-alpha, and MMP-1 and -3 for the primary analysis. The remaining cytokines will be examined in secondary analyses.

SECONDARY OUTCOMES:
To evaluate the reproducibility of cytokine assays in simultaneously collected blister fluid samples from normal patients. | study completion
To determine if there are differences within circulating and skin proteome and cytokine patterns between participants with cancer and healthy normal controls | study completion
To determine if cytokine levels and changes at the proteome level measured in blister fluid correlate with absorbed radiation skin dose, acute RTOG skin toxicity (>Grade 3), or late RTOG skin toxicity (>Grade 2). | study completion
To determine if changes in the proteome in blister fluid occur following exposure of the skin to low or high dose radiation | study completion
To determine how proteomic pattern changes in skin correlate with circulating proteomic patterns. | study completion
To determine how cytokine levels in skin correlate with circulating and urinary cytokine levels. | study completion

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Citrin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] D'Auria L, Pimpinelli F, Ferraro C, D'Ambrogio G, Giacalone B, Bellocci M, Ameglio F. Relationship between theoretical molecular weight and blister fluid/serum ratio of cytokines and five other molecules evaluated in patients with bullous pemphigoid. J Biol Regul Homeost Agents. 1998 Jul-Sep;12(3):76-80. PMID 9795835
- [Background] Riekki R, Parikka M, Jukkola A, Salo T, Risteli J, Oikarinen A. Increased expression of collagen types I and III in human skin as a consequence of radiotherapy. Arch Dermatol Res. 2002 Jul;294(4):178-84. doi: 10.1007/s00403-002-0306-2. Epub 2002 Apr 27. PMID 12111348
- [Background] Sonesson B, Rosengren E, Hansson AS, Hansson C. UVB-induced inflammation gives increased d-dopachrome tautomerase activity in blister fluid which correlates with macrophage migration inhibitory factor. Exp Dermatol. 2003 Jun;12(3):278-82. doi: 10.1034/j.1600-0625.2003.120307.x. PMID 12823441
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0120.html